CLINICAL TRIAL: NCT03026868
Title: Randomized Trails of Different Fixations for Acetabular Fracture Involving Quadrilateral Surface
Brief Title: Novel Quadrilateral Surface Plate for Acetabular Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZY2016
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-01

CONDITIONS: Fracture Dislocation
Keywords: acetabular; quadrilateral surface plate
MeSH Terms: conditions — Fracture Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- quadrilateral surface plate (Experimental): The fragments of the acetabulum were fixed with novel quadrilateral surface plate through Stoppa approach.
  Interventions: Procedure: quadrilateral surface plate

INTERVENTIONS:
Procedure: quadrilateral surface plate — Both anterior and posterior approaches were always conducted to manage the fragments of quadrilateral surface. Novel quadrilateral surface plate was used in this study to examine whether the fragments could be fixed through single Stoppa approach.

SUMMARY:
The novel plate could be used to manage acetabular fractures involving quadrilateral surface and posterior column, which may lower the intraoperative blood loss and reduce complication rate.

DETAILED DESCRIPTION:
Stoppa approach was more minimally invasive than ilioinguinal approach for pelvic and acetabular fractures. Then, Stoppa approach was widely used clinically. For the fragments involving quadrilateral surface, the Kocher-Langenbeck approach was added because the fixation of posterior fragments could not be obtained with reconstruction plate through single Stoppa approach. Novel quadrilateral surface plate was used in this study to examine its fixed role for posterior fragments. Functional outcome and complication were recorded to compare with the results treated with reconstruction plate. If good results were obtained for the patients fixed with quadrilateral surface plate, it was meaningful to popularize the fixed method.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Fracture involving quadrilateral surface
* Operation was conducted within 14 days
* Fixed with quadrilateral surface plate through Stoppa approach

Exclusion Criteria:

* Presented with a pathologic acetabular fracture
* Neuropathic arthropathy,dementia and other disease processes which made postoperative compliance unreliable
* Refused to participate
* Follow-up insufficient 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
fracture healing time | 4 months
  fracture line disappeared in the radiograph

SECONDARY OUTCOMES:
complication | 1 month
  wound infection, iatrogenic injury of vessels and nerves, nonunion

CONTACTS AND LOCATIONS:
Overall Officials: Ruipeng Zhang, M.D, Principal Investigator — Third Hospital of Hebei Medical University Department of Orthopaedic Surgery
Locations (1):
- Zhiyong Hou, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No